CLINICAL TRIAL: NCT05202951
Title: Status of Chronic Pain in Patients With Hemophilia.
Brief Title: Chronic Pain and Hemophilia
Acronym: HEMODOL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 LEBRETON 2; 2021-A01217-34 (Other: ANSM)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Hemophilia
Keywords: Chronic Pain; Hemophilia
MeSH Terms: conditions — Chronic Pain; Hemophilia A | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hemophilia: all adult patients follow-upin Hospital for hemophilia
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Electronic case report form integrating questionnaires on chronic pain related to haemophilia, associated-comorbidities, sociodemographic characteristics and analgesic treatments used.
  Other Names: RedCap web platform

SUMMARY:
Hemophilia (A and B) are X-linked hereditary bleeding disorders whose severity depends on the level of coagulation factor (FVIII or FIX respectively). Bleeding is mainly from joints (hemarthrosis) and muscles (hematoma). Nowadays, treatment is based on preventive or curative intravenous infusion of coagulation factor concentrates. Despite these treatments, there is joint deterioration that can be responsible for hemophilic arthropathy and chronic pain. This pain may be related to excess nociception during acute bleeding, but it may also be neuropathic. There are only a few studies that have looked at pain in hemophilia, but it is accepted that the vast majority of patients (especially those with severe forms) suffer from chronic pain. Because patients have become accustomed to this pain and physicians are still not very aware of how to assess it, this pain is not treated effectively.

In order to better manage pain in hemophilia, it is therefore necessary to characterize their pain and to know the nociceptive or neuropathic component. The aim of our study is therefore to study the prevalence, the nociceptive or neuropathic profile, the chronic aspect of pain and the main locations of pain in hemophilia. In addition to raising the awareness of physicians in the centers about pain management using specific questionnaires, this survey will help to better define chronic pain in hemophilia of all severities.

DETAILED DESCRIPTION:
This first French assessment of chronic pain in patients with haemophilia will permit to improve and generate new data about chronic pain related to haemophilia, associated-comorbidities, sociodemographic characteristics and analgesic treatments used.

These data will be retrieved using several questionnaires in the RedCap web plateform (eCRF).

The study will include 6 investigator centres and a minimum of 350 patients during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with haemophilia of any severity,
* Carrier female with low levels haemophilia (< 40%),
* ≥ 18 years of age and capable of giving informed consent to participate in research.

Exclusion Criteria:

* Patient's refusal to participate in the survey,
* Patient does not understand enough French (written and spoken) to complete the survey,
* Patient unable to complete the survey for logistical reasons (lack of internet access),
* Patient under protective measures (guardianship),
* Patients with known addictive comorbidities and/or cognitive disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of chronic pain disorders | through study completion, an average of 1 year
  Questionnaire "Brief Pain Inventory" (BPI) + History of chronic pain (≥ 3 months, Yes or No)

SECONDARY OUTCOMES:
Impact of chronic pain in daily life | through study completion, an average of 1 year
  Specific questions + Western Ontario and McMaster University Osteoarthritis (WOMAC)
Analgesic consumption | through study completion, an average of 1 year
  Type and quantity of analgesic used for treating chronic pain
Anxiodepressive disorders | through study completion, an average of 1 year
  Hospital Anxiety and Depression scale (HADS): this questionnaire makes it possible to detect anxiety and depressive disorders. It has 14 items sided from 0 to 3. Seven questions relate to anxiety and the 7 to the depressive dimension, thus obtaining two scores of up to 21.
Sleep disorders | through study completion, an average of 1 year
  MOS-Sleep scale (MOS-SS) questionnaire: this questionnaire deals with daytime sleepiness. It also looks at a person's ability to stay and fall asleep, how often they sleep and for how long, whether the sleep they get is adequate for their lifestyle, and any existing breathing factors that can affect sleep like sleep apnea.
Perceived injustice of chronic pain | through study completion, an average of 1 year
  Injustice Experience Questionnaire (IEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien LEBRETON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (10):
- France (10):
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen Normandie, Caen
  - CH Métropole Savoie, Chambéry
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CHU de LILLE, Lille
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de TOULOUSE, Toulouse